CLINICAL TRIAL: NCT03819816
Title: Development and Evaluation of an Application for Supporting Informal Caregivers of People With Dementia in Their Daily Life
Brief Title: Development and Evaluation of the DEA App
Acronym: DEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valentin Ritschl (Other)
Collaborators: FH Campus Wien, University of Applied Sciences (Other)
Responsible Party: Sponsor-Investigator, Valentin Ritschl, Principal Investigator, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DEA_APP_2019
Record Dates: First submitted 2019-01-23; First posted 2019-01-29 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Dementia
Keywords: informal caregivers; person with dementia; e-health solution
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEA-App (Experimental): The intervention (DEA) group will receive the newly developed app.
  Interventions: Other: DEA-App
- Standard Information group (Other): The control group will receive a leaflet on some general principles for promoting health and well-being in older adults with dementia.
  Interventions: Other: Standard Information group

INTERVENTIONS:
Other: DEA-App — The intervention (DEA) group will receive the newly developed app. DEA will consist of three simultaneous modules that provide multidimensional support for informal caregivers aiming to reduce the caregiver burden:
  1. Information module
     The information module consists of general information on the disease and the care of people suffering from dementia.
  2. Activity module
     The activity module suggests individualized activities and physical fitness exercises by a self-learning algorithm, which supports the caregiver to deliver more targeted and easier care.
  3. Communication module
  If two or more persons are caring for one person with dementia, the communication module provides a networking possibility.
  Arms: DEA-App
Other: Standard Information group — The control group will receive a leaflet on some general principles for promoting health and well-being in older adults with dementia.
  Arms: Standard Information group

SUMMARY:
Background, current situation, and motivation

According to current estimates, 100,000 people in Austria suffer from various types of dementia. According to forecasts, this number of people will rise to approximately 230,000 by 2050 due to the demographic development and the increase of the prevalence rate. Data from the service statistics show that 85% of dementia patients still live in the community in their homes and informal caregivers, such as relatives, support them. In total, more than 300,000 people care for their relatives in Austria in addition to professional support. However, not only the person affected from dementia suffers from the disease, but also, and often at a higher rate, the informal caregivers. Vice versa, the quality of life of those suffering from dementia is significantly influenced by the caregivers' competences and their strategies for resilience.

Study aim and hypothesis

The aim of this study is to evaluate the usability, acceptance, and effect of an app consisting of three modules that provide multidimensional support for informal caregivers of a person with dementia.

ELIGIBILITY:
Inclusion Criteria:

* informal caregivers of a person with dementia
* 18 years or older
* enough language skills to participate
* give written and oral informed consent
* have an Android smartphone or tablet (required to use the app).

Exclusion Criteria:

* none

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Burden Scale for Family Caregivers | 3 month after baseline
  The Burden Scale for Family Caregivers are rated on a scale from 0 (strongly disagree) to 3 (strongly agree). The score ranges from 0 to 84 points. Higher scores indicate greater caregiver burden

SECONDARY OUTCOMES:
12-item Short-Form Health Survey | 3 month after baseline
  The SF-12 is a shortened version of the 36-item Short Form Health Survey (SF-36). It is developed as an applicable instrument for measuring health-related quality of life.
Adult carers quality of life questionnaire | 3 month after baseline
  The Adult Carer Quality of Life Questionnaire is a simple instrument for use with adult carers. It measures quality of life in eight domains:
  1. support for caring,
  2. caring choice,
  3. caring stress,
  4. money matters,
  5. personal growth,
  6. sense of value,
  7. ability to care, and
  8. carer satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Tanja A Stamm, PhD, Principal Investigator — Medical University of Vienna
Locations (2):
- Austria (2):
  - Medical University of Vienna, Vienna
  - University of Applied Sciences FH Campus Wien, Vienna

IPD SHARING:
Plan to Share IPD: Undecided